CLINICAL TRIAL: NCT05009108
Title: Establishing of the Reliability of the Purdue Pegboard Test in Adults After a Stroke
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Rybářová, occupational therapist, Charles University, Czech Republic
Other Study IDs: 21/05/2021
Record Dates: First submitted 2021-08-12; First posted 2021-08-17 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Motor Activity
Keywords: Standardized test; Occupational therapy; Fine motor skills; Purdue Pegboard Test; Czech language; Inter-rater reliability; Internal variability; Stroke; Adults
MeSH Terms: conditions — Motor Activity; Stroke | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Czech adult patients after a stroke: Czech adults patients after a stroke will be asked to fill in a informed agreement and as well to answer short questionnaire. Then they will be tested by the Purdue Pegboard Test in only one session. Video of their performance will be obtained as well.
  Interventions: Diagnostic Test: Purdue Pegboard Test

INTERVENTIONS:
Diagnostic Test: Purdue Pegboard Test — At first, each person will be asked to fill in the informed agreement and answer short questionnaire. Than he/she will be tested by the Purdue Pegboard Test according to the Czech version of extended manuals for those tests in only one session. Audio recording of verbal instructions will be used and whole testing process will be video recorded which is necessary for establishing the internal variability and variability of results of the Purdue Pegboard Test.
  The results will be used only for establishing of the variability and inter-rater reliability of the Purdue Pegboard Test, not for patients' other interventions.
  Other Names: questionnaire

SUMMARY:
The main aim of the pilot project is to establish inter-rater reliability, internal variability and variability of results got by testing adults patients after a stroke by the use of Purdue Pegboard Test administered according to the new Czech extended version of its manual.

DETAILED DESCRIPTION:
New Czech manual for the Purdue Pegboard Test which is updated and extended by new rules for unification of their performing will be used for testing adult people with disability - adults after a stroke. The manuals include instructions for performing three trials of each subtest.

At least 30 adult patients after a stroke will be tested by use of Purdue Pegboard test administrated according to the new Czech extended version of its manual. Video of performance of each adult will be obtained. Performance of each patient, firstly in real time and secondly from video record will be evaluated twice, to obtain result for establishing all types of variability and reliability mentioned below.

The inter-rater reliability, internal variability and variability of results will be established.

ELIGIBILITY:
Inclusion Criteria:

* Czech language as a mother tongue
* age from 18 to 65 years
* patient after a stroke hospitalized at Rehabilitation institute Kladruby
* fine motor skills allowing them correct manipulation with components of Purdue Pegboard Test

Exclusion Criteria:

* severe disorder of orientation (neglect syndrome)
* use of drugs affecting attention
* vision impairment uncorrectable with glasses
* severe hearing loss
* inability to understand instructions
* inability to read or write
* inability to complete complete testing due to severe spasticity or spastic dystonia
* failure to sign Informed consent for probation with inclusion to research and Consent to the collection and processing of personal data during the study at the Rehabilitation institute Kladruby

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation
Study Population: Czech adult patients after a stroke
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
results from the Purdue Pegboard Test | 25 minutes
  number of parts put in the Pegboard according to the rules

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Rehabilitační ústav Kladruby, Kladruby
  - Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: No